CLINICAL TRIAL: NCT01506648
Title: Assessment of Zinc Absorption From a Phytic Acid Rich Complementary Food, Consumed by Young Children Immediately After the Addition of the Enzyme Phytase. A Randomized Single Blind Study
Brief Title: Assessment of Zinc Absorption From a Phytic Acid Rich Complementary Food
Status: Completed | Type: Observational
Sponsor: Swiss Federal Institute of Technology (Other)
Responsible Party: Principal Investigator, Prof. Michael B. Zimmermann, Prof, Swiss Federal Institute of Technology
Other Study IDs: INSTAPA-FP7-211484
Record Dates: First submitted 2012-01-09; First posted 2012-01-10 (Estimated); Last update posted 2016-11-28 (Estimated); Status verified 2016-11

CONDITIONS: Bioavailability

SUMMARY:
Assessment of zinc absorption from a phytic acid rich complementary food, consumed by young children immediately after the addition of the enzyme phytase. A randomized single blind study

ELIGIBILITY:
Inclusion Criteria:

1. 12-24 month old
2. Male of female
3. Height and weight between -2.0 SD and +2.0 SD with respect to WHO child growth standards.
4. No mineral and vitamin supplements 2 weeks prior to the study and during the whole duration of the study

Exclusion Criteria:

1. Body temperature ≥ 37.5°C
2. Hemoglobin ≤ 7g/dL
3. Positive RDT test
4. Any metabolic, gastrointestinal or chronic disease (according to the statement of the subject's parent) known chronic diseases at the gastrointestinal tract)
5. Long term mediation (that may affect zinc metabolism) during the whole study to interact with zinc metabolism (such as kidney diseases or

Ages: 12 Months to 24 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Study not related to a disease. Nutrition study without drug drug administration. Assessment of zinc absorption from a phytic acid rich complementary food, consumed by young children immediately after the addition of the enzyme phytase. A randomized single blind study
Sampling Method: Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2011-01; Primary Completion 2012-04 (Actual); Study Completion 2012-10 (Actual)

PRIMARY OUTCOMES:
Fractional absorption of zinc | 33 days
  Fractional absorption of zinc is estimated by using the double isotope tracer ratio technique by administering 67Zn as oral and 70Zn as intravenous stable isotopes.The urinary enrichment with both isotopes is measured in a spot urine sample by inductively coupled plasma mass spectrometry.

CONTACTS AND LOCATIONS:
Locations (1):
- CHU-Yalgado Ouédraogo, Service Pédiatrie, Ouagadougou, Burkina Faso